CLINICAL TRIAL: NCT07187375
Title: A Phase 2, Open-Label Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Pharmacodynamics of Crinecerfont in Pediatric Subjects 0 to <2 Years of Age With Congenital Adrenal Hyperplasia
Brief Title: Pharmacokinetics, Safety and Tolerability of Crinecerfont in Participants With Congenital Adrenal Hyperplasia Who Are Less Than 2 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-74788-CAH2011; 2024-514127-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; Crinecerfont
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — crinecerfont

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Crinecerfont (Experimental): Participants with CAH will receive crinecerfont during an initial 14-day treatment period, followed by an optional 36-month open-label extension (OLE).
  Interventions: Drug: Crinecerfont

INTERVENTIONS:
Drug: Crinecerfont — Oral solution

SUMMARY:
The main objective for this study is to evaluate the pharmacokinetics (PK) of crinecerfont in pediatric participants 0 to <2 years of age with congenital adrenal hyperplasia (CAH).

ELIGIBILITY:
Key Inclusion Criteria:

* Be a female or male between 0 to <2 years of age at screening.
* Have a medically confirmed diagnosis of classic CAH (salt wasting or simple virilizing) due to 21-hydroxylase deficiency (21-OHD).
* Be on a clinically stable regimen of hydrocortisone (and fludrocortisone, if applicable) treatment.

Key Exclusion Criteria:

* Have a known or suspected diagnosis of any of the other forms of classic CAH.
* Have any condition besides CAH that requires chronic daily therapy with orally administered steroids.
* Have any other clinically significant medical condition or chronic disease.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 0 Years to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-09-06 (Estimated); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Crinecerfont | Days 7 and 15

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Month 37

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Neurocrine Clinical Site, Berlin
  - Neurocrine Clinical Site, Heidelberg

IPD SHARING:
Plan to Share IPD: No